CLINICAL TRIAL: NCT06384859
Title: Effectiveness of Extracorporeal Shockwave Therapy Combined With Platelet-rich Plasma in the Treatment of Chronic Insertional Achilles Tendinopathy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pending
Record Dates: First submitted 2024-04-23; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Insertional Achilles Tendinopathy
Keywords: chronic insertional Achilles tendinopathy; extracorporeal shockwave therapy; platelet rich plasma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT + PRP (Experimental): Receive ESWT once a week for 4 weeks and PRP injection at a week later
  Interventions: Device: ESWT; Biological: PRP
- ESWT (Active Comparator): Receive ESWT once a week for 4 weeks
  Interventions: Device: ESWT

INTERVENTIONS:
Device: ESWT — Receive ESWT once a week for 4 weeks
Biological: PRP — Receive PRP injection at week 5
  Arms: ESWT + PRP

SUMMARY:
The goal of this clinical trial is to learn about the effectiveness of extracorporeal shockwave(ESWT) combined with platelet-rich plasma(PRP) to treat chronic insertional tendinopathy. The main questions it aims to answer are:

Does ESWT combined with PRP treatment reduce the symptom and improve functional score after treatment? What medical complication do participants have when receive the treatment?

Researchers will compare ESWT combined with PRP to ESWT treatment alone to see if ESWT combined with PRP works to treat chronic insertional tendinopathy.

Participants will:

* Receive ESWT once a week for 4 weeks then receive PRP injection at a week later or ESWT once a week for 4 weeks
* Visit the clinic at 6 weeks, 3 months, 6 months and 1 year after treatment for checkups and record functional score

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with insertional Achilles tendinopathy
* Had symptom more than 6 months
* Failed other standard conservative treatment (rest, medication, activity modification, stretching exercise, and heel lift orthosis)

Exclusion Criteria:

* Receive corticosteroid injection at the Achilles insertion
* History of infection around ankle and heel
* Has neurological deficit
* Has a contraindication for ESWT(hemophilia, coagulopathy or foot and ankle malignancy)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
VAS | 6 week, 3 months, 6 months and 1 year after treatment
  Visual Analogue Scale

SECONDARY OUTCOMES:
VAS-FA | 6 week, 3 months, 6 months and 1 year after treatment
  Visual analogue scale foot and ankle
FFI | 6 week, 3 months, 6 months and 1 year after treatment
  Foot functional index
FAAM | 6 week, 3 months, 6 months and 1 year after treatment
  Foot and Ankle Ability Measure

CONTACTS AND LOCATIONS:
Locations (1):
- Ramathibodi hospital, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code